CLINICAL TRIAL: NCT01701297
Title: The Effect of Probiotics on the Incidence of Spontaneous Bacterial Peritonitis in Patients With Cirrhosis and Ascites
Brief Title: VSL#3 and Spontaneous Bacterial Peritonitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to obtain QP release certification from the manufacturer (VSL3) for shipment of IMP
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: VSL Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10GA021; 2010-022886-92 (EudraCT Number); 10/H0405/81 (Other: NRES)
Record Dates: First submitted 2012-08-08; First posted 2012-10-05 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Decompensated Cirrhosis; Ascites
Keywords: Cirrhosis, ascites, infection
MeSH Terms: conditions — Ascites; Fibrosis; Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Co-trimoxazole (Active Comparator): Co-trimoxazole 960mg daily po
  Interventions: Drug: cotrimoxazole
- VSL#3 active (Experimental): VSL#3 active 2 sachets/daily
  Interventions: Drug: VSL#3 active
- VSL#3 placebo (Placebo Comparator): VSL#3 placebo 2 sachets/daily
  Interventions: Drug: VSL#3 placebo

INTERVENTIONS:
Drug: cotrimoxazole — Cotrimoxazole 960mg orally each day (two 480mg tablets)
  Other Names: Cotrimoxazole (septrin)
  Arms: Co-trimoxazole
Drug: VSL#3 active — The prescribed dose was 2 sachets (containing 900 billion bacteria) orally each day for 48 weeks
  Arms: VSL#3 active
Drug: VSL#3 placebo — This was two placebo sachets identical to VSL#3 active sachet. The prescribed dose was 2 sachets orally each day for 48 weeks
  Arms: VSL#3 placebo

SUMMARY:
Research question: Do oral probiotics in patients with cirrhosis and ascites reduce intestinal bacterial concentrations, ascitic bacterial DNA, SBP and bacteraemia compared to antibiotics or placebo?

This study is designed to investigate the effects of an oral probiotic (VSL#3; a mixture of "healthy" bacteria for the intestines) compared to an antibiotic or placebo in preventing infection developing in the abdominal fluid ("ascites") that collects in patients with advanced liver disease ("cirrhosis"). Patients already having had infection will be excluded from the study. Clear inclusion and exclusion criteria will be met and patients will be monitored throughout the study to examine whether they have required more hospitalisations, their rate infection in abdominal fluid or elsewhere and the level of liver function.

DETAILED DESCRIPTION:
The prevalence of cirrhosis is increasing in the UK. Decompensation heralds a poor outcome, with mortality in those developing ascites approximately 50% over the following 1-2 years. Spontaneous bacterial peritonitis (SBP) in ascitic fluid further reduces survival and occurs due to a combination of increased intestinal epithelial dysfunction, bacterial translocation to mesenteric lymph nodes and ascitic fluid, and reduced opsonisation and neutrophil function. Even with antibiotic treatment, 3-month mortality from SBP is approximately 40% and results in expensive in-patient care. Several studies have confirmed the benefit of secondary prophylaxis with long-term oral antibiotics in patients with advanced liver disease (e.g. norfloxacin, co-trimoxazole) and others suggest that in patients at high risk of developing SBP, primary antibiotic prophylaxis improves rates of sepsis and survival. Problems with these strategies include emergence of bacterial resistance, and development of antibiotic-associated diarrhoea (including C. difficile infection, which has a high case-fatality rate in those with cirrhosis). Local bacterial resistance profiles and association with C. difficile infection favour the choice of co-trimoxazole in our study population. Patients with advanced cirrhosis taking co-trimoxazole have previously demonstrated reduced liver-related outcomes such as infection and death3. Probiotic preparations alter intestinal bacterial flora and improve intestinal barrier and neutrophil function. Faecal bacterial counts of E. coli and Streptococcus (organisms commonly responsible for SBP) showed a 2-log fall with probiotics, although whether they could reduce the incidence of SBP remains unexamined.

ELIGIBILITY:
Inclusion criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with required disease/severity/symptoms as outlined in 6.3.1.
* Stable dose of current regular medication (e.g. diuretics, beta-blockers, vitamin supplementation) for at least 4 weeks prior to study entry.
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
* Participants have clinically acceptable laboratory tests and ECG within 14 days of enrolment.
* Able (in the Investigators opinion) and willing to comply with all study requirements.

Willing to allow their General Practitioner and consultant

Exclusion criteria:

* Female participants who is pregnant, lactating or planning pregnancy during the course of the study.
* Presence of hepatocellular carcinoma
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Participant who is terminally ill
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Use of antibiotics or probiotics in the last 2 weeks
* Known hypersensitivity to trimethoprim, sulphonamides or any other ingredients in co-trimoxazole tablet.
* History of acute porphyria or serious haematological disorder.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Liver-related mortality and liver related morbidity | 12 months

SECONDARY OUTCOMES:
Incidence of SBP, variceal bleeding, any non-SBP sepsis (e.g. pneumonia, urinary tract infection), clinical episodes of encephalopathy and the incidence of C. difficile infection. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin W James, BM BS FRCP PhD, Principal Investigator — NUH NHS Trust
Locations (1):
- NUH NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No